CLINICAL TRIAL: NCT05418439
Title: Study to Evaluate the Efficacy of Poppi Apple Cider Vinegar Prebiotic Soda to Improve Gut Health In Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drink Poppi (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20229 Poppi
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: bloating; abdominal pain; gassiness; heartburn
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Poppi ACV prebiotic soda (Experimental): Each day in the morning, for lunch, or in the afternoon, participants will drink one 12 fl oz. can of Poppi ACV prebiotic soda.
  Interventions: Dietary Supplement: Drink Poppi Soda

INTERVENTIONS:
Dietary Supplement: Drink Poppi Soda — Drink Poppi Vinager Soda

SUMMARY:
This exploratory observational trial provides the opportunity to gather information on the effect of daily consumption of Poppi Apple Cider Vinegar Prebiotic Soda on gut health and digestion.

DETAILED DESCRIPTION:
Individuals aged 18+ with a BMI under 30 and self-reported regular issues with IBS and/or poor digestion symptoms, including bloating, gassiness, heartburn, abdominal pain, constipation or associated symptoms (self-reported), but otherwise healthy will be chosen to participate in the study (see "4. Participant Definition"). Participants will be advised to discontinue any other oral supplement targeting the gut, including antibiotics, during the study and at least 3 months prior to.

Participants will be asked to complete the baseline survey on gut and skin health before the study starts.

Participants will also be asked to discontinue any additional soda consumption during the study.

Each day in the morning, for lunch, or in the afternoon, participants will drink one 12 fl oz. can of Poppi ACV prebiotic soda.

After 2 full weeks (day 14 of the study period) of drinking Poppi daily, participants will complete the 2-week follow up survey of gut and skin health.

After four weeks (day 28) of the study period, participants will complete the 4-week end-of-study follow up survey of gut and skin health. Making the whole study period four weeks.

The gut health surveys completed at baseline, week two and week four will be evaluated to determine the impact of Poppi ACV prebiotic soda on symptoms of poor gut health/digestion/IBS, including bloating, gas, heartburn, constipation and abdominal pain, as well as skin health.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45
* Male or Female
* Must be in generally good health
* BMI under 35
* Self-reported issues with gas, bloating, heartburn/acid reflux, abdominal pain or digestion
* Willing to maintain their standard dietary pattern, activity level and body weight for the duration of the study

Exclusion Criteria:

* Severe chronic conditions, including oncological conditions or psychiatric disease
* Currently pregnant, wanting to become pregnant, or breastfeeding for the duration of the study
* Taking any prescription medication targeting the gut
* Taking any supplements targeting the gut in the past month
* Use of antibiotics in the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in IBS symptoms [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale) of changes in IBS symptoms with higher scores representing an improved outcome.
Change in bowel movements [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale) of changes in stool frequency and consistency (constipation vs. diarrhea vs. normal) with higher scores representing an improved outcome.
Change in skin health [Time Frame: Baseline to 4 weeks) | 4 weeks
  Survey-based assessment (0-5 scale) of changes in perceived skin health with higher scores representing an improved outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No